CLINICAL TRIAL: NCT03233100
Title: FMT Treating Constipation Patients With Depression and/or Anxiety Symptoms - Clinical Efficacy and Potential Mechanisms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jianfeng Gong (Other)
Responsible Party: Sponsor-Investigator, Jianfeng Gong, Professor, Associate senior doctor, Jinling Hospital, China
Organization: Jinling Hospital, China (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STC-D-A-2017-FMT
Record Dates: First submitted 2017-07-22; First posted 2017-07-28 (Actual); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Constipation - Functional; Depressive Symptoms; Anxiety Symptoms; Gut-Brain Disorders
Keywords: FMT; gut microbiota; gut-brain disorder; constipation; depression; anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders; Constipation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FMT group (Experimental)
  Interventions: Other: FMT

INTERVENTIONS:
Other: FMT — fecal microbiota transplantation

SUMMARY:
Constipated patients often have mental problems such as depression and anxiety due to difficult defecation. Our previous studies have proved the efficacy of FMT treating constipation. Meanwhile it is believed that mental diseases are correlated to gut microbiota. This trial is based on the theory of the gut-brain-microbiota axis. Patients with constipation, depression and/or anxiety are performed FMT, laboratory, imaging and microbiota examinations, and clinical follow-up, to observe the clinical efficiency of FMT and the potential role of gut microbiome in these gut-brain disorders.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were diagnosed as functional constipation (FC) according to Rome Ⅳ criteria were enrolled.
* Age ≥ 18 years
* Body mass index of 18-25 kg/m2.
* HAMA ≥ 14 and/or HAMD (17 items) ≥ 17

Exclusion Criteria:

* History of sever mental disorders such as schizophrenia and bipolar disorder
* History of organic intestinal disorders
* History of gastrointestinal surgery
* Pregnant or breast-feeding women
* Infection with enteric pathogen
* Usage of probiotics, prebiotics, antibiotics within the last month
* Uncontrolled hepatic, renal, cardiovascular, and respiratory, or any diseases that in the opinion of the investigator, could affect intestinal transit and the intestinal microbiota.
* Patients who could not complete the follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-07-30 (Estimated); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
CSBMs per week | 12 weeks after treatment
  complete spontaneous bowl movements per week
HAMA | 12 weeks after treatment
  score of Hamilton Anxiety Rating Scale
HAMD | 12 weeks after treatment
  score of Hamilton Depression Rating Scale

SECONDARY OUTCOMES:
Wexner | pre, 2 weeks, 4 weeks, 8 weeks, 12weeks
  score of Wexner
PAC-SYM | pre, 2 weeks, 4 weeks, 8 weeks, 12weeks
  score of PAC-SYM
Bristol Bristol PAC-SYM | pre, 2 weeks, 4 weeks, 8 weeks, 12weeks
  score of Bristol score of Bristol
PAC-QOL | pre, 2 weeks, 4 weeks, 8 weeks, 12weeks
  score of PAC-QOL

OTHER OUTCOMES:
Gut microbiota analysis | pre, 4 weeks, 12 weeks
  Gut microbiota analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Generay Surgery, Jinling hosptal, Medical School of Nanjing University, Nanjing, Jiangsu, China